CLINICAL TRIAL: NCT03857477
Title: The BARCODE 1 Study: The Use of Genetic Profiling to Guide Prostate Cancer Targeted Screening.
Brief Title: The BARCODE 1 Study (Full Study): The Use of Genetic Profiling to Guide Prostate Cancer Targeted Screening.
Acronym: BARCODE1
Status: Active, not recruiting | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5044
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, blood, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stage 1: Caucasian men aged 55-69 to undergo genetic SNP profiling.
  Interventions: Genetic: Genetic SNP profiling
- Stage 2: Men from Stage 1 identified as having a higher genetic risk score (top 10%) for prostate cancer will be offered an MRI scan, prostate biopsy and prostate cancer screening.
  Interventions: Genetic: Genetic SNP profiling; Other: Prostate cancer screening; Procedure: MRI Scan; Procedure: Prostate biopsy

INTERVENTIONS:
Genetic: Genetic SNP profiling — Genetic SNP profiling of known prostate cancer predisposition SNPs will be performed on DNA extracted from saliva samples.
Other: Prostate cancer screening — Prostate cancer screening in the form of PSA testing will be offered to all men who have a benign biopsy result for five years in order to track development of cancer in the future.
  Groups: Stage 2
Procedure: MRI Scan — MRI scan will be offered to men identified within the top 10% genetic risk score profile.
  Other Names: MRI
  Groups: Stage 2
Procedure: Prostate biopsy — Transperineal prostate biopsy under local anaesthetic will be offered to men identified within the top 10% genetic risk score profile.
  Other Names: Transperineal Biopsy (TP biopsy)
  Groups: Stage 2

SUMMARY:
BARCODE 1 is a screening study designed to investigate the role of genetic profiling for targeting population prostate cancer screening. A pilot of 300 men were recruited aiming to inform the feasibility and accessibility of the study approach. The full study is an extension of the pilot study aiming to recruit a total of 5000 men.

DETAILED DESCRIPTION:
The BARCODE 1 study aims to evaluate genetic profiling using the known ~170 prostate cancer (PrCa) risk single-nucleotide polymorphisms (SNPs) as a means of offering targeted screening for PrCa in men at a genetically higher risk. Initially, 300 men were recruited via participating General Practices (GPs). The full study aimed to recruit an additional 4700 participants. Men aged 55-69 years who were likely to be eligible for the study were identified by GPs from medical records. Participants were contacted via invitation letters from GPs and if interested in the study were asked to sign a consent form and complete a questionnaire to confirm eligibility to participate. If eligible, men were then sent a DNA collection saliva kit. DNA from saliva was analysed with SNP profiling for the known ~170 clinically relevant SNPs. Men with a genetic risk equivalent to the top 10% of the population distribution (approximately 470 men in total from the full study) were invited for an MRI and a transperineal (TP) prostate biopsy under local anaesthetic (LA), plus further biological samples. Biopsy results will be correlated with the genetic score. The study also aims to determine the incidence and aggressiveness of prostate cancer in men within the top 10% of the genetic score. Furthermore, the association of MRI appearance and biological sample biomarker profile with prostate biopsy result in men at genetically higher prostate cancer risk undergoing targeted screening will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 55 to 69 years.
* Caucasian ethnicity.
* WHO performance status 0-2.
* Absence of any psychological, familial, sociological or geographical situation potentially hampering compliance with the study protocol and follow-up schedule.

Exclusion Criteria:

* Non-Caucasian ethnicity (including mixed race or Ashkenazi Jewish (excluded as these groups have different genetic risk profiles from those being studied).
* Previous diagnosis of cancer with a life-expectancy of less than five years.
* Negative prostate biopsy within one year before recruitment.
* Previous diagnosis of prostate cancer.
* Co-morbidities making prostate biopsy risk unacceptable (anticoagulants or antiplatelet medication including Warfarin, Clopidogrel, Apixaban, Dabigatran or other NOAC medications (Novel Oral Anti-Coagulant); poorly controlled diabetes, cardiovascular/respiratory disease, immunosuppressive medication or splenectomy).
* Men with body mass index (BMI) 40 and above.
* Men with BMI 35 and above plus other co-morbidities.
* Contraindications to having an MRI (pacemakers, aneurysm clips, metallic cardiac valve/stent, Ventriculo-Peritoneal (VP) shunt, cochlear implant, neurotransmitter, metallic foreign bodies in eye(s), other metalwork, claustrophobia).
* Any significant psychological conditions that may be worsened or exacerbated by participation in the study.

Ages: 55 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants must be of male gender at birth.
Study Population: Men of Caucasian ethnicity (not Mixed race or Jewish), aged 55 - 69 years, willing to undergo genetic SNP profiling.
Sampling Method: Non-Probability Sample
Enrollment: 4700 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Association of SNP genetic risk score with prostate biopsy results. | 5 years

SECONDARY OUTCOMES:
Incidence and aggressiveness of PrCa in men within the top 10% of the genetic score. | 5 years
Association of the biomarker profile with genetic score and biopsy results. | 5 years
Use of genetic profiling to target prostate cancer screening in a population screening clinical environment. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind A Eeles, FRCP, FRFR, Principal Investigator — Institute of Cancer Research and Royal Marsden Hospital
Locations (1):
- Institute of Cancer Research and Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data can be applied for via the Data Access Committee.

REFERENCES:
- [Background] McHugh JK, Bancroft EK, Saunders E, Brook MN, McGrowder E, Wakerell S, James D, Rageevakumar R, Benton B, Taylor N, Myhill K, Hogben M, Kinsella N, Sohaib AA, Cahill D, Hazell S, Withey SJ, Mcaddy N, Page EC, Osborne A, Benafif S, Jones AB, Patel D, Huang DY, Kaur K, Russell B, Nicholson R, Croft F, Sobczak J, McNally C, Mutch F, Bennett S, Kingston L, Karlsson Q, Dadaev T, Saya S, Merson S, Wood A, Dennis N, Hussain N, Thwaites A, Hussain S, Rafi I, Ferris M, Kumar P, James ND, Pashayan N, Kote-Jarai Z, Eeles RA; BARCODE1 Steering Committee and Collaborators. Assessment of a Polygenic Risk Score in Screening for Prostate Cancer. N Engl J Med. 2025 Apr 10;392(14):1406-1417. doi: 10.1056/NEJMoa2407934. PMID 40214032